CLINICAL TRIAL: NCT00753441
Title: Endoscopic Biliary Stenting on Demand Versus Surgical Biliary Bypass for Palliation of Patients With Advanced Cancer of the Pancreatic Head: STENTBY - A Randomized Controlled Trial
Brief Title: Endoscopic Stenting Versus Surgical Bypass for Low Bile Duct Obstruction by Cancer of the Pancreatic Head
Acronym: STENTBY
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low patient accrual
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Nuh Rahbari, MD, Heidelberg University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NNR-02
Record Dates: First submitted 2008-09-15; First posted 2008-09-16 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic cancer; Bile duct obstruction; Stent; Bypass
MeSH Terms: conditions — Pancreatic Neoplasms; Cholestasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Surgical bypass (choledochojejunostomy, in combination with gastroenterostomy if necessary)
  Interventions: Procedure: Surgical bypass
- B (Active Comparator): Endoscopic biliary stenting using metal stent (completed by duodenal stent, if necessary)
  Interventions: Procedure: Endoscopic stenting

INTERVENTIONS:
Procedure: Surgical bypass — Surgical bypass (choledochojejunostomy, in combination with gastroenterostomy if necessary)
  Arms: A
Procedure: Endoscopic stenting — Placement of a biliary metal stent (in combination with a duodenal metal stent in case of gastric outlet obstruction if necessary)
  Arms: B

SUMMARY:
The prognosis of patients with unresectable pancreatic cancer is dismal. Hence, palliation of tumor-associated symptoms, in particular jaundice due to low bile duct obstruction and gastric outlet obstruction, is the primary aim of these patients' care. Endoscopic stenting and surgical bypass are currently the two competing treatment options. There is currently no randomized trial comparing the recently developed metal stents to surgical bypass. Furthermore, there is very limited data on quality of life of these patients receiving either therapy. While endoscopic stenting represents the less invasive treatment, surgery may provide better long-term control requiring one-time treatment. Due to the incomplete evidence the present randomized controlled trial is designed to compare quality of life of patients undergoing endoscopic stenting on demand or surgical bypass for palliation of symptoms caused by cancer of the pancreatic head requiring with low bile duct obstruction.

ELIGIBILITY:
Inclusion Criteria:

* Age equal or greater than 18 years
* Diagnosis of unresectable cancer of the pancreatic head (after clinical, laboratory, radiological assessment) requiring palliative treatment for biliary obstruction. In unclear cases an exploratory laparotomy will be performed and resectability will be evaluated intraoperatively
* Operability certified by anesthesiologist
* Written informed consent

Exclusion Criteria:

* Intervention technically/medically not feasible
* Expected lack of compliance
* One treatment option considered to be clearly in favor of the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-02-01 (Actual); Primary Completion 2017-08-16 (Actual); Study Completion 2017-08-16 (Actual)

PRIMARY OUTCOMES:
Quality of life | 12 months
Serum bilirubin | 12 months

SECONDARY OUTCOMES:
Procedure-related complications | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Schmied, MD, Principal Investigator — Department of General, Visceral and Transplantation Surgery, University of Heidelberg
Locations (1):
- Universityhospital Heidelberg, Heidelberg, Germany